CLINICAL TRIAL: NCT01628159
Title: A Prospective, Multicenter, LEVANT 2 Continuation Registry of the Moxy™ Drug Coated Balloon for Treatment of Femoropopliteal Arteries
Brief Title: LEVANT 2 Continuation Registry of the Lutonix® Drug Coated Balloon (DCB)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL0002-09
Record Dates: First submitted 2012-06-19; First posted 2012-06-26 (Estimated); Results first posted 2020-04-10 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-03

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lutonix Drug Coated Balloon (Experimental): Formerly called the Moxy Drug Coated Balloon, the Lutonix Drug Coated Balloon (Lutonix DCB) is a paclitaxel coated balloon catheter
  Interventions: Device: Lutonix Drug Coated Balloon

INTERVENTIONS:
Device: Lutonix Drug Coated Balloon — balloon angioplasty with a drug coated balloon
  Other Names: Moxy Drug Coated Balloon

SUMMARY:
The purpose of the study is to collect additional safety and efficacy information on the Lutonix (formerly Moxy) Drug Coated Balloon for treatment of stenosis or occlusion of the femoral and popliteal arteries.

DETAILED DESCRIPTION:
The purpose of the study is to collect additional safety and efficacy information on the Lutonix (formerly Moxy) Drug Coated Balloon for treatment of stenosis or occlusion of the femoral and popliteal arteries through 5 years.

ELIGIBILITY:
Clinical Inclusion Criteria:

1. Male or non-pregnant female ≥18 years of age;
2. Rutherford Clinical Category 2-4;
3. Patient is willing to provide informed consent, is geographically stable and comply with the required follow up visits, testing schedule and medication regimen;

   Angiographic Lesion Inclusion Criteria:
4. Length ≤15 cm;
5. Up to two focal lesions or segments within the designated 15 cm length of vessel may be treated (e.g. two discrete segments, separated by several cm, but both falling within a composite length of <15 cm);
6. ≥70% stenosis by visual estimate;
7. Lesion location starts ≥1 cm below the common femoral bifurcation and terminates distally ≤2 cm below the tibial plateau AND ≥1 cm above the origin of the TP trunk;
8. de novo lesion(s) or non-stented restenotic lesion(s) >90 days from prior angioplasty procedure;
9. Lesion is located at least 3 cm from any stent, if target vessel was previously stented;
10. Target vessel diameter between ≥4 and ≤6 mm and able to be treated with available device size matrix;
11. Successful, uncomplicated (without use of a crossing device) antegrade wire crossing of lesion;
12. A patent inflow artery free from significant lesion (≥50% stenosis) as confirmed by angiography (treatment of target lesion acceptable after successful treatment of inflow artery lesions); NOTE: Successful inflow artery treatment is defined as attainment of residual diameter stenosis ≤30% without death or major vascular complication.
13. At least one patent native outflow artery to the ankle, free from significant (≥50%) stenosis as confirmed by angiography that has not previously been revascularized (treatment of outflow disease is NOT permitted during the index procedure);
14. Contralateral limb lesion(s) cannot be treated within 2 weeks before and/or planned 30 days after the protocol treatment in order to avoid confounding complications;
15. No other prior vascular interventions within 2 weeks before and/or planned 30 days after the protocol treatment.

Exclusion Criteria:

Patients will be excluded if ANY of the following conditions apply:

1. Pregnant or planning on becoming pregnant or men intending to father children;
2. Life expectancy of <5 years;
3. Patient is currently participating in an investigational drug or other device study or previously enrolled in this study; NOTE: Enrollment in another clinical trial during the follow up period is not allowed.
4. History of hemorrhagic stroke within 3 months;
5. Previous or planned surgical or interventional procedure within 2 weeks before or within 30 days after the index procedure;
6. History of MI, thrombolysis or angina within 2 weeks of enrollment;
7. Rutherford Class 0, 1, 5 or 6;
8. Renal failure or chronic kidney disease with MDRD GFR ≤30 ml/min per 1.73 m2 (or serum creatinine ≥2.5 mg/L within 30 days of index procedure or treated with dialysis);
9. Prior vascular surgery of the index limb, with the exception of remote common femoral patch angioplasty separated by at least 2 cm from the target lesion;
10. Inability to take required study medications or allergy to contrast that cannot be adequately managed with pre- and post-procedure medication;
11. Anticipated use of IIb/IIIa inhibitor prior to randomization;
12. Ipsilateral retrograde access;
13. Composite lesion length is >15 cm or there is no normal proximal arterial segment in which duplex flow velocity can be measured;
14. Significant inflow disease. Successful treatment of inflow disease allowed prior to target lesion treatment;
15. Known inadequate distal outflow (>50 % stenosis of distal popliteal and/or all three tibial vessels), or planned future treatment of vascular disease distal to the target lesion;
16. Sudden symptom onset, acute vessel occlusion, or acute or sub-acute thrombus in target vessel;
17. Severe calcification that renders the lesion un-dilatable;
18. Use of adjunctive treatment modalities (i.e. laser, atherectomy, cryoplasty, scoring/cutting balloon, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 657 (Actual)
Dates: Start 2012-06; Primary Completion 2018-09 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Rosenfield, MD, Principal Investigator — Massachusetts General Hospital; Prof. Dierk Scheinert, MD, Principal Investigator — University Leipzig
Locations (64):
- United States (39):
  - Good Samaritan Hospital, Los Angeles, California
  - North County Radiology Medial Group Inc., Oceanside, California
  - St. Joseph's Hospital, Orange, California
  - University of California Davis, Sacramento, California
  - Medical Center of the Rockies, Loveland, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - Washington Cardiology Center, Washington D.C., District of Columbia
  - Heart and Vascular Institute, Clearwater, Florida
  - Interventional Cardiolgists of Gainesville, Gainesville, Florida
  - Munroe Regional Medical Center, Ocala, Florida
  - Cardiovascular Associates, Elk Grove Village, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Edward Heart / Midwest Research Foundation, Oakbrook Terrace, Illinois
  - St. John's Hosptial, Springfield, Illinois
  - Allen County Cardiology, Fort Wayne, Indiana
  - St. Vincent Heart Center of Indianapolis, Indianapolis, Indiana
  - Promise Regional Medical Center, Hutchinson, Kansas
  - St. Francis Heart & Vascular Center, Topeka, Kansas
  - Massachusetts Genearl Hospital, Boston, Massachusetts
  - Detroit Medical Center, Detroit, Michigan
  - St. John's Hospital, Detroit, Michigan
  - Michigan Heart, Ypsilanti, Michigan
  - Mercy Hosptial, Coon Rapids, Minnesota
  - Forrest General Hospital, Hattiesburg, Mississippi
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Our Lady of Lourdes Medical Center, Cherry Hill, New Jersey
  - Mount Sinai Medical Center, New York, New York
  - Columbia Universtiy Medical Center, New York, New York
  - Wake Heart and Vascular, Raleigh, North Carolina
  - Christ Hospital / The Lindner Clinical Trial Center, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Mid Ohio Cardiology and Vascular Consultants, Columbus, Ohio
  - Jobst Vascular Institute, Toledo, Ohio
  - Univesrity of Toledo Medical Center, Toledo, Ohio
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Wellmont Cardiology Services, Kingsport, Tennessee
  - East Tennessee Heart Consultants, Knoxville, Tennessee
  - Austin Heart P.A., Austin, Texas
- Austria (2):
  - Medical University of Graz, Graz
  - Klinikum Klagenfurt, Klagenfurt
- Belgium (5):
  - OLV Ziekenhuis, Aalst
  - Imelda Ziekenhuis, Bonheiden
  - Flanders Medical Research Program, Dendermonde
  - Hospital Oost-Limburg, Genk
  - Ghent University Hospital, Ghent
- Germany (15):
  - Herz-Zentrum, Bad Krozingen
  - Jewish Hospital, Berlin
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Diakonissenanstalt zu Flensburg, Flensburg
  - Hamburg University Cardiovascular Center, Hamburg
  - University Clinical Center Heidelberg, Heidelberg
  - Herz-Und Gefasszentrum, Immenstadt im Allgäu
  - Practice for Interventional Radiology, Kaiserslautern
  - Westpfalz Clinic, Kusen
  - University Leipzig, Leipzig
  - University Magdeburg, Magdeburg
  - University of Munich, Munich
  - Universtiy Clinic Muenster, Münster
  - Ernst von Bergham Clinic, Potstdam
  - University of Tübingen, Tübingen
- Switzerland (3):
  - University Hospital, Bern
  - Canton Hospital Lucerne, Lucerne
  - University Hospital, Zurich, Zurich

IPD SHARING:
Plan to Share IPD: No
Not at this time.

REFERENCES:
- [Derived] Ouriel K, Adelman MA, Rosenfield K, Scheinert D, Brodmann M, Pena C, Geraghty P, Lee A, White R, Clair DG. Safety of Paclitaxel-Coated Balloon Angioplasty for Femoropopliteal Peripheral Artery Disease. JACC Cardiovasc Interv. 2019 Dec 23;12(24):2515-2524. doi: 10.1016/j.jcin.2019.08.025. Epub 2019 Sep 28. PMID 31575518

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lutonix Drug Coated Balloon
Started | 657
Completed | 493
Not Completed | 164

BASELINE CHARACTERISTICS:
Arm/Group | Lutonix Drug Coated Balloon
Number analyzed (Participants) | 657
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.7 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 238
  Male | 419
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 645
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 657
Baseline Rutherford Classification [Count of Participants; unit: Participants] — Rutherford Classification is on an ascending scale from 0 to 6. Lower classifications on the scale indicate more favorable outcomes.
  0 - Asymptomatic
  1. - Mild claudication
  2. - Moderate claudication
  3. - Severe claudication
  4. - Rest pain
  5. - Ischemic ulceration not exceeding ulcer of the digits of the foot
  6. - Sever ischemic ulcers or frank gangrene
  Participants
    Rutherford 0 | 0
    Rutherford 1 | 0
    Rutherford 2 | 240
    Rutherford 3 | 379
    Rutherford 4 | 38
    Rutherford 5 | 0
    Rutherford 6 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Unanticipated Device- or Drug- Related Adverse Events Through 60 Months Post Index Procedure
Time Frame: 60 months Post Index Procedure
Measure: Number; unit: Events
Arm/Group | Lutonix Drug Coated Balloon
Number analyzed (Participants) | 657
Events | 0

2. Secondary Outcome: Number of Patients With Freedom From All-Cause Perioperative (≤ 30 Day) Death and Freedom From Index Limb Amputation, Index Limb Re-Intervention, and Index-Limb-Related Death at 1, 6, 12, 24, 36, 48, and 60 Months Post Index Procedure
Description: Composite of freedom from all-cause perioperative (≤ 30 day) death and freedom from the following at 1, 6, 12, 24, 36, 48, and 60 months: index limb amputation, index limb re-intervention, and index-limb-related death.
Time Frame: 1, 6, 12, 24, 36, 48 and 60 months Post Index Procedure
Population: The number of participants (n) varies from the total number of participants (N) in the study as n depends on the number of participants for which data was available at the given time-point analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Lutonix Drug Coated Balloon
Number analyzed (Participants) | 657
Participants
  1 Month Post Index Procedure | 638
  6 months post-index procedure: number analyzed (Participants) | 633
  6 months post-index procedure | 596
  12 months post Index procedure: number analyzed (Participants) | 623
  12 months post Index procedure | 525
  24 Months Post Index Procedure: number analyzed (Participants) | 592
  24 Months Post Index Procedure | 434
  36 Months Post Index Procedure: number analyzed (Participants) | 568
  36 Months Post Index Procedure | 385
  48 Months Post Index Procedure: number analyzed (Participants) | 547
  48 Months Post Index Procedure | 347
  60 Months Post Index Procedure: number analyzed (Participants) | 529
  60 Months Post Index Procedure | 320

3. Secondary Outcome: Number of Acute Device Success at Time of Index Procedure
Description: In certain procedures, more than one device was use resulting in a higher number of devices (894) than participants (657) for this endpoint.
Time Frame: At time of Index Procedure
Measure: Count of Units; unit: Devices
Units Other Than Participants: Devices
Arm/Group | Lutonix Drug Coated Balloon
Number analyzed (Participants) | 657
Number analyzed (Devices) | 894
Devices | 894

4. Secondary Outcome: Number of Participants With Freedom From All-cause Death, Index Limb Amputation Above the Ankle and Target Vessel Revascularization (TVR) at 30 Days Post Index Procedure
Description: This VIVA Safety Endpoint is defined as Freedom at 30 days from all-cause death, index limb amputation above the ankle and target vessel revascularization (TVR).
Time Frame: 30 days post index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Lutonix Drug Coated Balloon
Number analyzed (Participants) | 647
Participants | 642

5. Secondary Outcome: Number of Participants With Freedom From Index Limb Amputation, Index Limb Re-Intervention, and Index-Limb-Related Death at 1, 6, 12, 24, 36, 48, and 60 Months Post Index Procedure (PPI)
Time Frame: 1, 6, 12, 24, 36, 48, and 60 months post index procedure
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Lutonix Drug Coated Balloon
Number analyzed (Participants) | 657
Participants
  Death : 1 month PPI: number analyzed (Participants) | 647
  Death : 1 month PPI | 1
  Death : 6 months PPI: number analyzed (Participants) | 636
  Death : 6 months PPI | 4
  Death : 12 months PPI: number analyzed (Participants) | 626
  Death : 12 months PPI | 8
  Death : 24 months PPI: number analyzed (Participants) | 601
  Death : 24 months PPI | 21
  Death : 36 months PPI: number analyzed (Participants) | 592
  Death : 36 months PPI | 45
  Death : 48 months PPI: number analyzed (Participants) | 585
  Death : 48 months PPI | 67
  Death : 60 months PPI: number analyzed (Participants) | 573
  Death : 60 months PPI | 83
  Major Amputation : 1 month PPI: number analyzed (Participants) | 646
  Major Amputation : 1 month PPI | 0
  Major Amputation : 6 months PPI: number analyzed (Participants) | 632
  Major Amputation : 6 months PPI | 0
  Major Amputation : 12 months PPI: number analyzed (Participants) | 620
  Major Amputation : 12 months PPI | 0
  Major Amputation : 24 months PPI: number analyzed (Participants) | 585
  Major Amputation : 24 months PPI | 1
  Major Amputation : 36 months PPI: number analyzed (Participants) | 557
  Major Amputation : 36 months PPI | 2
  Major Amputation : 48 months PPI: number analyzed (Participants) | 524
  Major Amputation : 48 months PPI | 4
  Major Amputation : 60 months PPI: number analyzed (Participants) | 495
  Major Amputation : 60 months PPI | 6
  Minor Amputation : 1 month PPI: number analyzed (Participants) | 646
  Minor Amputation : 1 month PPI | 1
  Minor Amputation : 6 months PPI: number analyzed (Participants) | 632
  Minor Amputation : 6 months PPI | 1
  Minor Amputation : 12 months PPI: number analyzed (Participants) | 620
  Minor Amputation : 12 months PPI | 1
  Minor Amputation : 24 months PPI: number analyzed (Participants) | 584
  Minor Amputation : 24 months PPI | 2
  Minor Amputation : 36 months PPI: number analyzed (Participants) | 556
  Minor Amputation : 36 months PPI | 3
  Minor Amputation : 48 months PPI: number analyzed (Participants) | 523
  Minor Amputation : 48 months PPI | 6
  Minor Amputation : 60 months PPI: number analyzed (Participants) | 493
  Minor Amputation : 60 months PPI | 6
  Amputation Free Survival 1 month PPI: number analyzed (Participants) | 647
  Amputation Free Survival 1 month PPI | 646
  Amputation Free Survival : 6 months PPI: number analyzed (Participants) | 636
  Amputation Free Survival : 6 months PPI | 632
  Amputation Free Survival : 12 months PPI: number analyzed (Participants) | 626
  Amputation Free Survival : 12 months PPI | 618
  Amputation Free Survival : 24 months PPI: number analyzed (Participants) | 602
  Amputation Free Survival : 24 months PPI | 580
  Amputation Free Survival : 36 months PPI: number analyzed (Participants) | 593
  Amputation Free Survival : 36 months PPI | 547
  Amputation Free Survival : 48 months PPI: number analyzed (Participants) | 585
  Amputation Free Survival : 48 months PPI | 515
  Amputation Free Survival : 60 months PPI: number analyzed (Participants) | 575
  Amputation Free Survival : 60 months PPI | 487
  Total TLR : 1 month PPI: number analyzed (Participants) | 646
  Total TLR : 1 month PPI | 3
  Total TLR : 6 months PPI: number analyzed (Participants) | 632
  Total TLR : 6 months PPI | 21
  Total TLR : 12 months PPI: number analyzed (Participants) | 621
  Total TLR : 12 months PPI | 78
  Total TLR : 24 months PPI: number analyzed (Participants) | 589
  Total TLR : 24 months PPI | 133
  Total TLR : 36 months PPI: number analyzed (Participants) | 565
  Total TLR : 36 months PPI | 154
  Total TLR : 48 months PPI: number analyzed (Participants) | 540
  Total TLR : 48 months PPI | 168
  Total TLR : 60 months PPI: number analyzed (Participants) | 520
  Total TLR : 60 months PPI | 174
  Total TVR : 1 month PPI: number analyzed (Participants) | 646
  Total TVR : 1 month PPI | 4
  Total TVR : 6 months PPI: number analyzed (Participants) | 632
  Total TVR : 6 months PPI | 26
  Total TVR : 12 months PPI: number analyzed (Participants) | 621
  Total TVR : 12 months PPI | 83
  Total TVR : 24 months PPI: number analyzed (Participants) | 589
  Total TVR : 24 months PPI | 144
  Total TVR : 36 months PPI: number analyzed (Participants) | 565
  Total TVR : 36 months PPI | 167
  Total TVR : 48 months PPI: number analyzed (Participants) | 542
  Total TVR : 48 months PPI | 184
  Total TVR : 60 months PPI: number analyzed (Participants) | 523
  Total TVR : 60 months PPI | 192
  Reintervention Thrombosis1 month PPI: number analyzed (Participants) | 646
  Reintervention Thrombosis1 month PPI | 0
  Reintervention Thrombosis : 6 months PPI: number analyzed (Participants) | 632
  Reintervention Thrombosis : 6 months PPI | 0
  ReinterventionThrombosis : 12 months PPI: number analyzed (Participants) | 620
  ReinterventionThrombosis : 12 months PPI | 1
  Reintervention Thrombosis : 24 months PPI: number analyzed (Participants) | 584
  Reintervention Thrombosis : 24 months PPI | 3
  ReinterventionThrombosis : 36 months PPI: number analyzed (Participants) | 557
  ReinterventionThrombosis : 36 months PPI | 4
  Reintervention Thrombosis : 48 months PPI: number analyzed (Participants) | 523
  Reintervention Thrombosis : 48 months PPI | 4
  ReinterventionThrombosis : 60 months PPI: number analyzed (Participants) | 494
  ReinterventionThrombosis : 60 months PPI | 5
  Cardiovascular Hospitalization : 1 month PPI: number analyzed (Participants) | 647
  Cardiovascular Hospitalization : 1 month PPI | 5
  Cardiovascular Hospitalization : 6 months PPI: number analyzed (Participants) | 634
  Cardiovascular Hospitalization : 6 months PPI | 33
  Cardiovascular Hospitalization : 12 months PPI: number analyzed (Participants) | 623
  Cardiovascular Hospitalization : 12 months PPI | 57
  Cardiovascular Hospitalization : 24 months PPI: number analyzed (Participants) | 592
  Cardiovascular Hospitalization : 24 months PPI | 60
  Cardiovascular Hospitalization : 36 months PPI: number analyzed (Participants) | 565
  Cardiovascular Hospitalization : 36 months PPI | 60
  Cardiovascular Hospitalization : 48 months PPI: number analyzed (Participants) | 533
  Cardiovascular Hospitalization : 48 months PPI | 60
  Cardiovascular Hospitalization : 60 months PPI: number analyzed (Participants) | 506
  Cardiovascular Hospitalization : 60 months PPI | 60
  Major Vascular Complication : 1 month PPI: number analyzed (Participants) | 648
  Major Vascular Complication : 1 month PPI | 12
  Major Vascular Complication : 6 months PPI: number analyzed (Participants) | 635
  Major Vascular Complication : 6 months PPI | 20
  Major Vascular Complication : 12 months PPI: number analyzed (Participants) | 623
  Major Vascular Complication : 12 months PPI | 29
  Major Vascular Complication : 24 months PPI: number analyzed (Participants) | 592
  Major Vascular Complication : 24 months PPI | 47
  Major Vascular Complication : 36 months PPI: number analyzed (Participants) | 567
  Major Vascular Complication : 36 months PPI | 51
  Major Vascular Complication : 48 months PPI: number analyzed (Participants) | 539
  Major Vascular Complication : 48 months PPI | 53
  Major Vascular Complication : 60 months PPI: number analyzed (Participants) | 513
  Major Vascular Complication : 60 months PPI | 54

6. Secondary Outcome: Number of Participants With Technical and Procedural Success
Time Frame: At time of index procedure
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Lutonix Drug Coated Balloon
Number analyzed (Participants) | 657
Participants
  Technical Success: number analyzed (Participants) | 644
  Technical Success | 566
  Procedural Success: number analyzed (Participants) | 644
  Procedural Success | 565

7. Secondary Outcome: Number of Participants With Primary Patency of the Target at 6, 12, and 24 Months Post Index Procedure
Description: Primary patency is defined as freedom from target lesion restenosis by core lab adjudication (DUS ≥ 2.5) and target lesion revascularization (TLR).
Time Frame: 6, 12, and 24 months post index procedure
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Lutonix Drug Coated Balloon
Number analyzed (Participants) | 657
Participants
  6 months post index procedure: number analyzed (Participants) | 590
  6 months post index procedure | 483
  12 months post index procedure: number analyzed (Participants) | 583
  12 months post index procedure | 386
  24 months post index procedure: number analyzed (Participants) | 547
  24 months post index procedure | 298

8. Secondary Outcome: Change From Baseline of Index-limb Resting Ankle Brachial Index (ABI) at 6, 12, and 24 Months Post Index Procedure
Description: Presented is a summary of the Mean change in resting Ankle Brachial Index (ABI) from baseline through 24 months post index procedure. The ABI is defined as a ratio of ankle to brachial (upper arm) artery systolic blood pressure and aims at determining how well the blood is flowing in the legs. A lower ABI number suggests more Peripheral Arterial Disease.
Time Frame: 6, 12, and 24 months post index procedure
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | Lutonix Drug Coated Balloon
Number analyzed (Participants) | 657
Index
  6 months post index procedure: number analyzed (Participants) | 572
  6 months post index procedure | 0.19 (0.27)
  12 months post index procedure: number analyzed (Participants) | 545
  12 months post index procedure | 0.18 (0.27)
  At 24 months post index procedure: number analyzed (Participants) | 484
  At 24 months post index procedure | 0.16 (0.28)

9. Secondary Outcome: Number of Participants With Freedom From Target Lesion Revascularization (TLR) at 1, 6, 12, and 24 Months Post Index Procedure
Time Frame: 1, 6, 12, and 24 months post index procedure
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Lutonix Drug Coated Balloon
Number analyzed (Participants) | 657
Participants
  1 month post index procedure: number analyzed (Participants) | 646
  1 month post index procedure | 643
  6 months post index procedure: number analyzed (Participants) | 632
  6 months post index procedure | 611
  12 months post index procedure: number analyzed (Participants) | 621
  12 months post index procedure | 543
  24 months post index proceedure: number analyzed (Participants) | 589
  24 months post index proceedure | 456

10. Secondary Outcome: Improvement From Baseline in Rutherford Classification (Index Limb) at 6, 12, and 24 Months Post Index Procedure
Description: The endpoint summarizes the change in index-limb Rutherford Classification of participants from baseline through 24 months. Data is presented as shift from baseline Rutherford Classification data using the following categories: 1) Improvement, 2) Same, and 3) Worsened.
Time Frame: 6, 12, and 24 months post index procedure
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Lutonix Drug Coated Balloon
Number analyzed (Participants) | 657
Participants
  6 months from baseline: number analyzed (Participants) | 611
  6 months from baseline: Improved | 540
  6 months from baseline: Same | 49
  6 months from baseline: Worsened | 22
  12 months from baseline: number analyzed (Participants) | 581
  12 months from baseline: Improved | 498
  12 months from baseline: Same | 62
  12 months from baseline: Worsened | 21
  24 months from baseline: number analyzed (Participants) | 536
  24 months from baseline: Improved | 459
  24 months from baseline: Same | 57
  24 months from baseline: Worsened | 20

11. Secondary Outcome: Number of Participants With Primary Patency Based on Alternative Peak Systolic Velocity Ratio (PSVR) Thresholds at 6, 12, and 24 Months Post Index Procedure
Description: * Alternative Primary and Secondary Patency based on alternative definitions of Duplex Ultrasonography (DUS) Peak Systolic Velocity Ratio (PSVR) <2.0 and <3.0
  * Duplex Ultrasonography (DUS) Clinical Patency (DUS Peak Systolic Velocity Ratio (PSVR) <2.5 without prior Clinically Driven TLR)
Time Frame: 6, 12, and 24 months post index procedure
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Lutonix Drug Coated Balloon
Number analyzed (Participants) | 657
Participants
  DUS PSVR >= 3.0 : 6 months post index procedure: number analyzed (Participants) | 479
  DUS PSVR >= 3.0 : 6 months post index procedure | 411
  DUS PSVR >= 3.0 : 12 months post index procedure: number analyzed (Participants) | 457
  DUS PSVR >= 3.0 : 12 months post index procedure | 295
  DUS PSVR >= 3.0 : 24 months post index procdure: number analyzed (Participants) | 427
  DUS PSVR >= 3.0 : 24 months post index procdure | 213
  DUS PSVR >= 2.5 : 6 months post index procedure: number analyzed (Participants) | 475
  DUS PSVR >= 2.5 : 6 months post index procedure | 396
  DUS PSVR >= 2.5 : 12 months post index procedure: number analyzed (Participants) | 462
  DUS PSVR >= 2.5 : 12 months post index procedure | 289
  DUS PSVR >= 2.5 : 24 months post index procdure: number analyzed (Participants) | 432
  DUS PSVR >= 2.5 : 24 months post index procdure | 203
  DUS PSVR >= 2.0 : 6 months post index procedure: number analyzed (Participants) | 476
  DUS PSVR >= 2.0 : 6 months post index procedure | 345
  DUS PSVR >= 2.0 : 12 months post index procedure: number analyzed (Participants) | 466
  DUS PSVR >= 2.0 : 12 months post index procedure | 242
  DUS PSVR >= 2.0 : 24 months post index procdure: number analyzed (Participants) | 454
  DUS PSVR >= 2.0 : 24 months post index procdure | 176

ADVERSE EVENTS:
Time Frame: From Post Index Procedure to End of Follow up Period (5-Year visit window).
Description: All Serious Adverse Events (SAE) presented in table were CEC-Adjudicated as probably or highly probably device-related.
  All non-serious Adverse Events (AE) presented in AE table are site reported and not all may be device-related events.
  The number of participants affected by non-serious events (528 out of 657 participants) is for all AEs reported in study, not only for events over the 5% threshold.
Arm/Group | Lutonix Drug Coated Balloon
All-Cause Mortality (participants affected / at risk) | 83/657
Serious Adverse Events (participants affected / at risk) | 67/657
Other Adverse Events (participants affected / at risk) | 528/657
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lutonix Drug Coated Balloon (N=657)
Infection, local (Infections and infestations) | 1 (1)
Infection (systemic) (Infections and infestations) | 1 (1) — Infection (systemic) requiring antibiotics.
Significant hemorrhage (General disorders) | 1 (1) — Access site: Significant hemorrhagic event requiring transfusion.
Pseudoaneurysm (Vascular disorders) | 1 (1) — Access site: Pseudoaneurysm
Target vessel injury (Vascular disorders) | 21 (21) — Angiographic event: Target vessel injury:/dissection with study treatment.
Distal embolization with study treatment (Vascular disorders) | 3 (3) — Angiographic event.
Distal embolization with post treatment (Vascular disorders) | 1 (1) — Angiographic event
Clot/Thrombus formation (Vascular disorders) | 1 (1) — Angiographic event: Thrombosis.
Other angiographic event (Vascular disorders) | 1 (1) — Events in this category were not collected in a way that allows their separation into specific categories or by specific events terms.
Restenosis of study lesion (Vascular disorders) | 3 (3) — Vascular event
Clinically-driven Target Lesion Revascularization (Vascular disorders) | 26 (26) — Vascular event: Clinically-driven target (study) lesion revascularization (TLR)
Target (study) vessel revascularization (TVR) (Vascular disorders) | 2 (2) — Vascular event
Target (study) limb ishchemia (Vascular disorders) | 1 (1) — Vascular event
Other vascular event (Vascular disorders) | 1 (1) — Not specified. Events in this category were not collected in a way that allows their separation into specific categories or by specific events terms.
Claudication (Vascular disorders) | 11 (11) — Vascular event
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lutonix Drug Coated Balloon (N=657)
Arrhytmia (Cardiac disorders) | 34 (36)
Hypertension (Cardiac disorders) | 43 (50)
Other cardiovascular events (Cardiac disorders) | 67 (87) — Cardiovascular events, not specified. Events in this category were not collected in a way that allows their separation into specific categories or by specific events terms.
Gastrointestinal events (other) (Gastrointestinal disorders) | 79 (128) — Gastrointestinal events, not specified. Events in this category were not collected in a way that allows their separation into specific categories or by specific events terms.
Local Infection (Infections and infestations) | 52 (69)
Neurological events (other) (Nervous system disorders) | 54 (64) — Events in this category were not collected in a way that allows their separation into specific categories or by specific events terms.
Respiratory (other) (Respiratory, thoracic and mediastinal disorders) | 52 (67) — Events in this category were not collected in a way that allows their separation into specific categories or by specific events terms.
Back pain (Musculoskeletal and connective tissue disorders) | 67 (72)
Claudication (Musculoskeletal and connective tissue disorders) | 55 (59)
Skeletal, spine and muscular events (Other) (Musculoskeletal and connective tissue disorders) | 155 (241) — Events in this category were not collected in a way that allows their separation into specific categories or by specific events terms.
Restenosis (Vascular disorders) | 35 (36) — Target Lesion: Restenosis event.
Renal failure/ insufficiency (Renal and urinary disorders) | 35 (37) — Genito-urinary system event.
Urinary infection (Renal and urinary disorders) | 46 (65) — Genito-urinary system event.
Various (General disorders) | 241 (527) — Not otherwise described. Events in this category were not collected in a way that allows their separation into specific categories or by specific events terms.
Vessel specific events (Other) (General disorders) | 41 (44) — Vessel specific events in the leg (not target lesion or target vessel). Events in this category were not collected in a way that allows their separation into specific categories or by specific events terms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-03-26): https://cdn.clinicaltrials.gov/large-docs/59/NCT01628159/Prot_SAP_000.pdf